CLINICAL TRIAL: NCT01506414
Title: A Multicentre Investigation of Recombinant Human Thrombopoietin (Rh-TPO) Combine With Low-dose Rituximab in Management of Steroid-Resistant/Relapsed Immune Thrombocytopenia (ITP)
Brief Title: Recombinant Human Thrombopoietin in Combination With Rituximab in Immune Thrombocytopenia (ITP)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ming Hou (Other)
Collaborators: Peking Union Medical College Hospital (Other); Chinese Academy of Medical Sciences (Other); First Affiliated Hospital, Sun Yat-Sen University (Other); West China Hospital (Other); Shandong Provincial Hospital (Other Government); Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other); Zhejiang University (Other)
Responsible Party: Sponsor-Investigator, Ming Hou, Director of Hematology Department, Shandong University
Organization: Shandong University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ITP-003
Record Dates: First submitted 2011-11-16; First posted 2012-01-10 (Estimated); Last update posted 2016-04-20 (Estimated); Status verified 2012-01

CONDITIONS: Purpura; Idiopathic Thrombocytopenic Purpura
Keywords: Purpura; Idiopathic Thrombocytopenic Purpura
MeSH Terms: conditions — Purpura; Purpura, Thrombocytopenic, Idiopathic | interventions — Rituximab; Thrombopoietin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- combination treatment (Experimental)
  Interventions: Drug: rhTPO in combination with Rituximab

INTERVENTIONS:
Drug: rhTPO in combination with Rituximab — Rituximab was given intravenously at a dose of 100 mg weekly for 4 consecutive weeks (Day 1, 8, 15, 22). Rh-TPO (TPIAOTM, a product of Sunshine Pharmaceutical Co Ltd, China, approved by China State Food and Drug Administration) was given subcutaneously at a dose of 1.0 μg/kg（300u/kg）for 14 days (Day 1-14).
  Other Names: Recombinant Human Thrombopoietin; Recombinant Human TPO; rhTPO combine with Rituximab; Recombinant Human Thrombopoietin combine with Rituximab; Recombinant Human TPO combine with Rituximab

SUMMARY:
The purpose of this study is to determine whether Recombinant Human Thrombopoietin (rh-TPO) in combination with Rituximab are effective and safe in the management of Steroid-Resistant/Relapsed Immune Thrombocytopenia (ITP).

DETAILED DESCRIPTION:
Rituximab was given intravenously at a dose of 100 mg weekly for 4 consecutive weeks (Day 1, 8, 15, 22). Rh-TPO (TPIAOTM, a product of Sunshine Pharmaceutical Co Ltd, China, approved by China State Food and Drug Administration) was given subcutaneously at a dose of 1.0 μg/kg（300u/kg）for 14 days (Day 1-14). Platelet count (PC) was monitored every three or four days until day 22, followed by tests every week. Platelet transfusion was administered to patients with active bleeding symptoms or to those whose PC<10×10^9/L. Patients were followed for 3 months, and any adverse effects were recorded during the period of treatment and during the follow-up.

ELIGIBILITY:
Inclusion Criteria:

1. Meet the diagnostic criteria for immune thrombocytopenia.
2. Untreated hospitalized patients, may be male or female, between the ages of 18 ~ 80 years.
3. To show a platelet count <30×10^9/L, and with bleeding manifestations.
4. Willing and able to sign written informed consent.

Exclusion Criteria:

1. Received chemotherapy or anticoagulants or other drugs affecting the platelet counts within 3 months before the screening visit.
2. Received second-line ITP-specific treatments (eg, cyclophosphamide, 6-mercaptopurine, vincristine, vinblastine, etc) within 3 months before the screening visit.
3. Received high-dose steroids or IVIG in the 3 weeks prior to the start of the study.
4. Current HIV infection or hepatitis B virus or hepatitis C virus infections.
5. Severe medical condition (lung, hepatic or renal disorder) other than chronic ITP. Unstable or uncontrolled disease or condition related to or impacting cardiac function (e.g., unstable angina, congestive heart failure, uncontrolled hypertension or cardiac arrhythmia)
6. Female patients who are nursing or pregnant, who may be pregnant, or who contemplate pregnancy during the study period.
7. Have a known diagnosis of other autoimmune diseases, established in the medical history and laboratory findings with positive results for the determination of antinuclear antibodies, anti-cardiolipin antibodies, lupus anticoagulant or direct Coombs test.
8. Patients who are deemed unsuitable for the study by the investigator.

Ages: 16 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 91 (Actual)
Dates: Start 2009-06; Primary Completion 2013-08 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Evaluation of platelet response (Complete Response) | The time frame is up to 3 months per subject
  CR. A complete response (CR) was defined as a sustained (≥ 3 months) platelet count ≥ 100×10^9/L without recurrence of thrombocytopenia
Evaluation of platelet response (R) | The time frame is up to 3 months per subject
  R. A response (R) was defined as a sustained (≥ 3 months) platelet count ≥ 30×10^9/L without recurrence of thrombocytopenia
Evaluation of platelet response (No Response) | The time frame is up to 3 months per subject
  NR.No response (NR) was defined as platelet count < 30 × 10^9/L or a less than two fold increase in platelet count from baseline or the presence of bleeding. Platelet count must be measured on two occasions more than a day apart.

SECONDARY OUTCOMES:
The number and frequency of therapy associated adverse events | up to 3 months per subject

CONTACTS AND LOCATIONS:
Overall Officials: Hou Ming, Dr., Principal Investigator — Shandong University
Locations (1):
- Qilu Hospital, Shandong University, Jinan, Shandong, China

REFERENCES:
- [Background] Provan D, Stasi R, Newland AC, Blanchette VS, Bolton-Maggs P, Bussel JB, Chong BH, Cines DB, Gernsheimer TB, Godeau B, Grainger J, Greer I, Hunt BJ, Imbach PA, Lyons G, McMillan R, Rodeghiero F, Sanz MA, Tarantino M, Watson S, Young J, Kuter DJ. International consensus report on the investigation and management of primary immune thrombocytopenia. Blood. 2010 Jan 14;115(2):168-86. doi: 10.1182/blood-2009-06-225565. Epub 2009 Oct 21. PMID 19846889
- [Background] Rodeghiero F, Stasi R, Gernsheimer T, Michel M, Provan D, Arnold DM, Bussel JB, Cines DB, Chong BH, Cooper N, Godeau B, Lechner K, Mazzucconi MG, McMillan R, Sanz MA, Imbach P, Blanchette V, Kuhne T, Ruggeri M, George JN. Standardization of terminology, definitions and outcome criteria in immune thrombocytopenic purpura of adults and children: report from an international working group. Blood. 2009 Mar 12;113(11):2386-93. doi: 10.1182/blood-2008-07-162503. Epub 2008 Nov 12. PMID 19005182
- [Background] Cheng Y, Wong RS, Soo YO, Chui CH, Lau FY, Chan NP, Wong WS, Cheng G. Initial treatment of immune thrombocytopenic purpura with high-dose dexamethasone. N Engl J Med. 2003 Aug 28;349(9):831-6. doi: 10.1056/NEJMoa030254. PMID 12944568
- [Background] Mazzucconi MG, Fazi P, Bernasconi S, De Rossi G, Leone G, Gugliotta L, Vianelli N, Avvisati G, Rodeghiero F, Amendola A, Baronci C, Carbone C, Quattrin S, Fioritoni G, D'Alfonso G, Mandelli F; Gruppo Italiano Malattie EMatologiche dell'Adulto (GIMEMA) Thrombocytopenia Working Party. Therapy with high-dose dexamethasone (HD-DXM) in previously untreated patients affected by idiopathic thrombocytopenic purpura: a GIMEMA experience. Blood. 2007 Feb 15;109(4):1401-7. doi: 10.1182/blood-2005-12-015222. Epub 2006 Oct 31. PMID 17077333